CLINICAL TRIAL: NCT05100212
Title: Umbilical or Adult Donor Red Blood Cells to Transfuse Extremely Low Gestational Age Neonates. A Randomized Trial to Assess the Effect on Retinopathy of Prematurity Severity.
Brief Title: umBilical Or Adult Donor Red Blood Cells in Extremely Low Gestational Age Neonates and Retinopathy of Prematurity (BORN)
Acronym: BORN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4364
Record Dates: First submitted 2021-10-14; First posted 2021-10-29 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-10

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Intervention Model Description: Interventional, randomized, controlled, double-blind, with an adaptive design to evaluate safety and efficacy of allogeneic CB-RBC transfusions.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adult-RBC transfusions (Active Comparator): Adult-red blood cell concentrate transfusions
  Interventions: Biological: adult donor RBC concentrates
- CB-RBC transfusions (Experimental): Cord blood-red blood cell concentrate transfusions
  Interventions: Biological: cord blood-RBC concentrates

INTERVENTIONS:
Biological: cord blood-RBC concentrates — Patients in the experimental arm are candidates to receive CB-RBC units until the completion of 29 weeks of postmenstrual age (29+6). In case of unavailability of an ABO/Rh matched CB-RBC unit, patients receive adult -RBC (standard transfusions).
  Other Names: cord blood packed RBC
  Arms: CB-RBC transfusions
Biological: adult donor RBC concentrates — Patients in the comparator arm are candidates to receive adult donor-RBC units
  Other Names: adult donor packed RBC
  Arms: Adult-RBC transfusions

SUMMARY:
Extremely low gestational age neonates (ELGAN, i.e., born before 28 gestation weeks) are among the most heavily transfused pediatric patients. In this clinical setting, repeated red blood cell (RBC) transfusions independently predict a poor outcome, with a higher risk for mortality and morbidity. Recent studies from our own and other groups highlighted a close association between low levels of fetal hemoglobin (HbF) and severity of retinopathy of prematurity (ROP) and bronchopulmonary dysplasia (BPD), two disabilities that frequently complicate preterm birth. This association is not surprising, considering that 1) preterm neonates have a highly immature antioxidant reserve and both ROP and BPD rely on the oxidative damage as underlying mechanism; 2) in comparison with HbA, HbF is endowed with higher oxygen affinity, greater redox potential, higher tetrameric stability, and higher ability to generate unbound nitric oxide, all functions potentially protective in presence of an oxidative challenge; 3) in normal prenatal life, developing organ and tissues are exposed exclusively to HbF until last weeks of gestation; 4) in preterm neonates, the switch of the synthesis from HbF to HbA occurs around their due date, i.e., several weeks after the premature birth; 5) when preterm neonates receive transfusions, their tissues are abruptly exposed to high levels of HbA. We have recently run a pilot trial demonstrating as a proof-of-concept that transfusing cord blood red blood cell concentrates (CB-RBC) effectively prevents or restrains the HbF loss consequent to adult donor standard transfusions (A-RBC). This study explores the hypothesis that transfusing CB-RBCs instead of A-RBC may lower the incidence of severe ROP in ELGANs needing transfusions.

ELIGIBILITY:
Inclusion Criteria:

* gestational age (GA) at birth between 24+0 and 27+6 weeks
* signed informed consent of parents.

Exclusion Criteria:

One or more of the following:

* maternal-fetal immunization
* hydrops fetalis
* major congenital malformations associated or not with genetic syndromes
* previous transfusions
* hemorrhage at birth
* congenital infections
* health care team deeming it inappropriate to approach the infant's family for informed consent.

Ages: 24 Weeks to 27 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Retinopathy of prematurity | up to the age of 40 weeks
  Incidence of severe ROP (stage 3 and higher) in CB-RBC and A-RBC arms

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Teofili, MD, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (10):
- Italy (10):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo,, Foggia
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Evangelico Villa Betania, Naples
  - AORN Santobono-Pausilipon, Napoli
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Fondazione Policlinico Universitario A.Gemelli IRCCS, Rome
  - Città della Salute e della Scienza, Torino

REFERENCES:
- [Derived] Teofili L, Papacci P, Dani C, Cresi F, Remaschi G, Pellegrino C, Bianchi M, Ansaldi G, Campagnoli MF, Vania B, Lepore D, Franco FGS, Fabbri M, de Vera d' Aragona RP, Molisso A, Beccastrini E, Dragonetti A, Orazi L, Pasciuto T, Mozzetta I, Baldascino A, Locatelli E, Valentini CG, Giannantonio C, Carducci B, Gabbriellini S, Albiani R, Ciabatti E, Nicolotti N, Baroni S, Mazzoni A, Besso FG, Serrao F, Purcaro V, Coscia A, Pizzolo R, Raffaeli G, Villa S, Mondello I, Trimarchi A, Beccia F, Ghirardello S, Vento G. Cord blood transfusions in extremely low gestational age neonates to reduce severe retinopathy of prematurity: results of a prespecified interim analysis of the randomized BORN trial. Ital J Pediatr. 2024 Aug 7;50(1):142. doi: 10.1186/s13052-024-01714-w. PMID 39113069
- [Derived] Teofili L, Papacci P, Orlando N, Bianchi M, Pasciuto T, Mozzetta I, Palluzzi F, Giaco L, Giannantonio C, Remaschi G, Santosuosso M, Beccastrini E, Fabbri M, Valentini CG, Bonfini T, Cloclite E, Accorsi P, Dragonetti A, Cresi F, Ansaldi G, Raffaeli G, Villa S, Pucci G, Mondello I, Santodirocco M, Ghirardello S, Vento G. BORN study: a multicenter randomized trial investigating cord blood red blood cell transfusions to reduce the severity of retinopathy of prematurity in extremely low gestational age neonates. Trials. 2022 Dec 13;23(1):1010. doi: 10.1186/s13063-022-06949-8. PMID 36514106